CLINICAL TRIAL: NCT06446947
Title: Identification de Marqueurs de Mauvais Pronostic Clinique du Sepsis Par Analyse épigénétique.
Brief Title: Identification of Markers of Poor Clinical Prognosis in Sepsis by Epigenetic Analysis
Acronym: EPISEPSIS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM23_0006
Record Dates: First submitted 2024-05-29; First posted 2024-06-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Sepsis Syndrome; Septic Shock; Sepsis
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Shock, Septic; Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and RNA extracted from patient blood samples will be preserved during the study. At the end of the analysis, the remaining samples will be discarded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic shock: Patients with sepsis admitted to intensive care who developed septic shock.
  Interventions: Other: blood sampling
- No septic shock: Patients with sepsis admitted to critical care with a favorable outcome (no septic shock)
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Blood sampling (6ml) on admission and a second on discharge from intensive care.

SUMMARY:
Sepsis is a multifactorial syndrome characterized by a dynamic course and a clinical outcome dependent on several factors, and responsible for one in five deaths worldwide. The aim of this trial is to identify new prognostic markers for the progression of sepsis to septic shock, by comparing epigenetic markers between patients who have or have not developed severe forms of sepsis.

The main objective of this preliminary study is to identify prognostic markers for the progression of sepsis to septic shock, i.e. to compare targeted markers between subjects with sepsis who progress to septic shock versus subjects with sepsis who do not progress to septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Male patients,
* Patients between 45 and 75 years of age,
* Patients undergoing major esophageal or digestive carcinological surgery,
* Patients with post-operative gram-negative bacterial sepsis (proven or suspected in the context of organ failure).

Exclusion Criteria:

* patients under 45 and aged 76 and over,
* female patients,
* non-carcinological or minor surgery,
* non-esophageal or non-digestive surgery,
* Gram-positive bacterial or fungal infections in the absence of associated BGN,
* patients with hematological cancer,
* immunocompromised patients,
* septic surgery (surgical site infection),
* patients expressing opposition to data collection and analysis (clinical and/or biological) within the regulatory framework of the study,
* patients under guardianship or curatorship,
* patients not affiliated to a social security system or equivalent in France,
* patients deprived of their liberty.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients admitted to critical care for sepsis after thoracic or chest surgery.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Identify prognostic markers for the progression of sepsis to septic shock | 18 months
  Compare targeted markers between subjects with sepsis progressing to septic shock versus subjects with sepsis not progressing to septic shock.

SECONDARY OUTCOMES:
Epigenetic markers comparaison | 18 months
  Epigenetic markers and associated candidate genes identified in PBMC at the time of sepsis between the group of subjects progressing to septic shock and the group of subjects not progressing to septic shock.
Differentials in epigenetic marks and associated candidate genes | 18 months
  Compare differentials in epigenetic marks and associated candidate genes (sepsis, second sampling) between the group of subjects progressing to septic shock and the group of subjects not progressing to septic shock
Epigenetic marks and associated candidate genes identified in PBMC | 18 months
  In both groups, compare the epigenetic marks and associated candidate genes identified in PBMC during sepsis with those identified in PBMC collected at the time of septic shock or discharge from critical care.

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Service Anesthésie Réanimation - Hôpital Nord - Assistance Publique Hôpitaux de Marseille, Marseille, Bouches du Rhône, France

IPD SHARING:
Plan to Share IPD: No